CLINICAL TRIAL: NCT00731913
Title: A Randomized, Prospective Trial Evaluating Surgeon-Preference in Selection of Absorbable Suture Material
Brief Title: A Comparison of Monosyn and Monocryl Sutures in Surgical Wounds
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Gary Rogers, Tufts Medical Center
Other Study IDs: 8229
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Wounds
Keywords: Surgical wounds; Sutures
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound | interventions — glycolide E-caprolactone copolymer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Subjects with skin lesions requiring surgical excision and repair. One half of the each wound received Monocryl suture and the other half received Monosyn suture.
  Interventions: Other: Absorable, monofilament sutures: Monosyn and Monocryl
- 2: Subjects with skin lesions requiring surgical excision and repair. One half of the each wound received Monocryl suture and the other half received Monosyn suture.
  Interventions: Other: Absorable, monofilament sutures: Monosyn and Monocryl

INTERVENTIONS:
Other: Absorable, monofilament sutures: Monosyn and Monocryl — Subjects were randomized to Monosyn vs. Monocryl suture arms. The designated skin lesion was removed surgically. The surgical repair of the defect was performed by dividing the wound in half by a single Prolene suture. The appropriate suture was opened by the Study Coordinator and passed sterilely to the surgical technician. The surgical technician loaded the suture, and passed it in a blinded fashion to the physician who closed the appropriate half of the surgical defect. One half of the wound was closed with one suture and the other half was closed with the other suture. Each patient served as their own control, as both sutures were used in each study patient.
  Other Names: Monofilament, absorbable sutures

SUMMARY:
To better understand surgeon preference when using synthetic, absorbable, monofilament suture by comparing two similar appearing FDA-approved sutures, Monosyn (Aesculap) and Monocryl (Ethicon).

DETAILED DESCRIPTION:
Physicians have used suture to close wounds for at least 4,000 years. Archaeological records from ancient Egypt show that Egyptians used linen and animal sinew to close wounds. In ancient India, physicians used the pincers of beetles or ants to staple wounds shut. They then cut the insects' bodies off, leaving their jaws (staples) in place. Other natural materials used to close wounds include flax, hair, grass, cotton, silk, pig bristles, and animal gut.

The fundamental principles of wound closure have changed little over 4,000 years. Successful closure of wound involves surgical techniques coupled with knowledge of the physical characteristics and handling of the suture and needle. The selection of proper suture material in closing any surgical defect is important in wound healing, minimizing infection, and achieving optimal cosmetic and functional results.

A great deal of progress has been made since Egyptian times with regard to suture materials and manufacturing processes. Today, sutures are available with a wide variety of characteristics, configuration, manipulability, coefficient of friction, solubility, strength, and immunogenic properties. Yet, sutures are currently rather crudely classified based on a numeric scale according to diameter and tensile strength; descending from 10 to 1, and then descending again from 1-0 to 12-0. This study aims to explore the factors that are important to a surgeon when choosing sutures via evaluating surgeon preference for two types of synthetic, absorbable, monofilament sutures: Monosyn and Monocryl. We hope to initiate a more nuanced exploration of how suture characteristics influence surgeon preference, beyond filament type and size, and how makers of suture may better report and represent these factors.

ELIGIBILITY:
Inclusion Criteria:

* Specific eligibility requirements included surgical defects that are linear, without curvature, 3.0 cm in length or greater and extending into the subcutis or fascia.
* All surgical defects were required to be closed primarily (that is without flaps or grafts) and had equal skin integrity on both halves of their surgical defects.
* All subjects were capable of providing written informed consent.

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with skin lesions requiring surgical removal were eligible for our study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
subjective surgeon preference for both suture types. | 2 weeks

SECONDARY OUTCOMES:
Objective handling characteristics as major determinants of surgeon preference for the sutures. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Rogers, MD, Principal Investigator — Tufts Medical Center; Linh K. Lu, MD, PhD, Study Director — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States